CLINICAL TRIAL: NCT00132236
Title: Smoking Cessation of Patients With COPD: A Multi-Center, Randomized, Placebo Controlled Nurse Conducted Smoking Cessation Trial
Brief Title: Nurse Smoking Cessation of Patients With Chronic Obstructive Pulmonary Disease (COPD) With Nicotine Replacement Therapy (NRT) and Behavioral Support
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KA01096gms; CTN980-CHC-9015-027
Record Dates: First submitted 2005-08-17; First posted 2005-08-19 (Estimated); Last update posted 2005-10-21 (Estimated); Status verified 2005-07

CONDITIONS: Smoking; COPD
Keywords: smoking cessation; nicotine sublingual tablets; behaviour support; smoking reduction; quality of life; COPD; weight
MeSH Terms: conditions — Smoking; Pulmonary Disease, Chronic Obstructive; Smoking Cessation; Smoking Reduction; Body Weight

INTERVENTIONS:
Drug: nicotine sublingual tablets
Behavioral: low and high behavior support

SUMMARY:
This is a smoking cessation study with COPD patients where the researchers wanted to evaluate if nicotine sublingual tablets or placebo combined with low or high individual support could increase ½ and 1 year quit rates.

DETAILED DESCRIPTION:
Placebo, controlled, randomized, double-blind trial with 400-1000 smoking COPD patients with FEV-1 < 90 % predicted normal with the use of nicotine sublingual nicotine tablets or placebo for 12 weeks combined with individual clinic visits with low or high intensity conducted by trained nurses in several centres in pulmonary clinics in Denmark. Outcome was smoking cessation and smoking reduction after ½ and 1 year as self declared smoking status confirmed by carbon monoxide in expired air< 10 ppm. Secondary outcomes were change in body-weight, quality of life (SF-36 and SGRQ), symptoms, lung function, adverse events.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients (FEV1/FVC<70% and FEV1<90 % predicted)
* Smoking 1 cigarette daily or more
* Willing to follow the protocol

Exclusion Criteria:

* Used NRT or bupropion the last week
* Not able or willing to adhere to the protocol
* Estimated survival < 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2002-02; Study Completion 2004-06

PRIMARY OUTCOMES:
smoking cessation after 6 and 12 months

SECONDARY OUTCOMES:
smoking reduction after 12 months
change in quality of life (St. George Respiratory Questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Tønnesen, M.D., Ph.D., Study Chair — Pulm. dept. Gentofte University Hospital
Locations (7):
- Denmark (7):
  - Dept. pulm. medicine, Århus kommunehospital, Aarhus
  - Dept. pulm. medicine, Bispebjerg Hospital, Copenhagen
  - Dept of Pulm. medicine, Helsingør Sygehus, Elsinore
  - Pulm. Dept., Frederiksberg Hospital, Frederiksberg, Copenhagen
  - Pulm. Dept, Gentofte University Hospital, Hellerup
  - Dept. pulm. medicine, Nykøbing Falster Sygehus, Nykøbing Falster
  - Pulm. dept, Odense University Hospital, Odense